CLINICAL TRIAL: NCT06908850
Title: Erogenous Zones in Adult Males After Complete Spinal Cord Injury
Brief Title: The Aim of This Research is to Better Understand How Complete Spinal Cord Injury May Change Erogenous Zones in Adult Males
Acronym: QualiEroSCI
Status: Enrolling by invitation | Type: Observational
Sponsor: Fondation Garches (Other)
Responsible Party: Principal Investigator, Nadine Streit, PHD student, Fondation Garches
Other Study IDs: QualiEroSCI
Record Dates: First submitted 2025-03-20; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury; Spinal Cord Injury No Sensory/Motor in S4-S5
Keywords: Sexuality; Erogenous zones; Men; Semi-structured interviews
MeSH Terms: conditions — Spinal Cord Injuries; Sexuality; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A complete spinal cord injury (SCI) in men is characterized by the total loss of motor skills and sensations below the injury. The loss of penile sensation, the erogenous zone primarily involved in sexual response, is involved in sexual dysfunction, impacting sexual pleasure and quality of life. The management of genito-sexual dysfunction is a priority for paraplegic patients, ahead of bladder-sphincter and motor functions. For tetraplegic patients, the restoration of genito-sexual functions is their second priority after the upper limb motor skills recovery (Anderson, 2004)(Anderson et al., 2007). Medical assistance is currently available to i) restore erectile function allowing penetrative sexual intercourse, ii) enable sperm collection for reproductive purposes, iii) assisted reproductive techniques which allowing most often these patients to achieve their fatherhood goals (Giuliano et al., 2019)(Chochina et al., 2016)(Lombardi et al., 2015). Nevertheless, the assessment and management of the loss of genital sensations have been poorly studied, alike sexual pleasure and satisfaction in SCI patients (Philpott et al., 2006).

Erogenous zones are regions of the body that elicit sexual pleasure and trigger or enhance sexual arousal when appropriately stimulated. The discovery of other forms of physical intimacy that move away from the traditional scripts of phallo-centric male sexuality (Earle et al., 2020)(Giurleo et al., 2022)(Ostrander, 2009)(Burns et al., 2008) could improve sexual pleasure. The stimulation of hypersensitive regions in the skin areas corresponding to the lesion level and above has the potential to represent one of the strategies to compensate the lack of sensitivity of the genital-sexual organs (Hohmann, 1972)(Bach-y-Rita, 1999)(Elliott, 2002)(Anderson et al., 2007)(Lopez et al., 2008)(Alexander & Marson, 2018). But again, these data are scares and limited to few testimonials.

The aim of the present research program is to identify, define and characterize erogenous zones in men with complete SCI in the absence of sensitivity of the genitals.

The study design is a qualitative observational study, and the consolidated criteria for reporting qualitative research (COREQ) will be followed (Tong et al., 2007). A minimum of fourteen semi-structured interviews with men with a complete SCI followed in a neuro-urology department will be conducted with the recruitment stopped once data saturation is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Complete spinal cord injury
* Heterosexual
* Sexual activity prior to the injury

Exclusion Criteria:

* Syringomyelia
* Other neurological condition
* No sexual activity since the injury

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: heterosexual adult men with a complete spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
Caracterization of the erogenous zones | At the time of the interview (Baseline)
  Semi structured interviews to identifie the phenomenology behind the erogenous zones
Localization of the erogenous zones | At the time of the interview (Baseline)
  Body map chart

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Raymond Poincaré, Garches, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chochina L, Naudet F, Chehensse C, Manunta A, Damphousse M, Bonan I, Giuliano F. Intracavernous Injections in Spinal Cord Injured Men With Erectile Dysfunction, a Systematic Review and Meta-Analysis. Sex Med Rev. 2016 Jul;4(3):257-269. doi: 10.1016/j.sxmr.2016.02.005. Epub 2016 Mar 29. PMID 27871959
- [Background] Bach-y-Rita P, W Kercel S. Sensory substitution and the human-machine interface. Trends Cogn Sci. 2003 Dec;7(12):541-6. doi: 10.1016/j.tics.2003.10.013. PMID 14643370
- [Background] Anderson KD, Borisoff JF, Johnson RD, Stiens SA, Elliott SL. Long-term effects of spinal cord injury on sexual function in men: implications for neuroplasticity. Spinal Cord. 2007 May;45(5):338-48. doi: 10.1038/sj.sc.3101978. Epub 2006 Oct 10. PMID 17016492
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] Alexander MS, Marson L. The neurologic control of arousal and orgasm with specific attention to spinal cord lesions: Integrating preclinical and clinical sciences. Auton Neurosci. 2018 Jan;209:90-99. doi: 10.1016/j.autneu.2017.01.005. Epub 2017 Jan 25. PMID 28222972